CLINICAL TRIAL: NCT02546752
Title: Use of a Patient Education/Messaging Platform to Increase Uptake and Series Completion of the HPV Vaccine
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Regenstrief Institute, Inc. (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Merck - 20
Record Dates: First submitted 2015-09-09; First posted 2015-09-11 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Human Papilloma Virus Infection Type 11; Human Papilloma Virus Infection Type 16; Human Papilloma Virus Infection Type 18; Human Papilloma Virus Infection Type 6; Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- THEO Video Arm (Experimental): THEO is interactive patient engagement software that runs on an iPad tablet platform (developed by Noble.MD). Two programs have been developed. Parents/guardians of children who have not received the first HPV vaccine, will first assess whether the family has already decided in favor of the HPV vaccine or if they would like more information. The parent/guardian will be shown a video specific to where they are in the decision-making process. After completion, the THEO system will then ask the parent/guardian a series of Post Video questions. Parents/guardians of children who have received the first or second vaccine in the series, will emphasize the need to make the first vaccine "count". Pre and post video questions have been developed.
  Interventions: Other: THEO
- Usual Care Arm (No Intervention): This arm will receive usual care.

INTERVENTIONS:
Other: THEO — THEO is interactive patient engagement software that runs on an iPad tablet platform (developed by Noble.MD). THEO is the intervention in this study.
  Arms: THEO Video Arm

SUMMARY:
This primary goal of this study is to assess whether patient whose parents watch a standardized digital video using the integrated digital approach during a routine office visit are more likely to accept a dose of HPV vaccine (1st, 2nd, or 3rd dose) compared to those not completing the program. The study team anticipates eligible patients in the intervention clinics to have higher rates of HPV vaccine acceptance (1st, 2nd, or 3rd doses) than patients in the usual care comparison clinics.

Additionally, the study team is interested in determining the impact of the integrated system on clinical workflow by measuring the number of minutes of each patient office visit when using the system compared to the number of minutes of each visit in offices where the system is not used.

Although this is a descriptive/exploratory aim, our expectation is that the THEO system will have minimal impact on patient flow.

DETAILED DESCRIPTION:
Brief Summary of Design: This is a 2-arm randomized study, with randomization occurring at the level of clinic. Five clinics will be included (2 implementing the THEO video; 3 providing usual care). All five clinics have been using the Child Health Improvement through Computer Automation System (CHICA) for several years. The evaluation phase of the study will last for approximately 6-7 months.

The CHICA System

The Child Health Improvement through Computer Automation system (CHICA) is a computer based decision support system that operates as a front end to the electronic medical record system (EMR). When a child is registered in the clinic, the registration system sends an HL7 ADT (registration) message to CHICA. In response, CHICA requests a download of the patient's record from the EMR. CHICA applies a rule base consisting of hundreds of Arden Syntax rules to the data in the record to select 20 yes/no questions that are displayed on an electronic tablet. The family answers the questions and returns the tablet to the medical assistant who enters the child's height, weight and other measurements onto another page on the tablet.

At the same time that CHICA produces the questions for family, it sends an HL7 request to CHIRP, the Indiana immunization registry. In response, CHICA receives a download of the child's immunization record. The download includes CHIRP's "forecast" of the immunizations for which the patient is due.

At the end of these processes, CHICA produces several paper documents. The first is the physician worksheet (PWS). The PWS includes up to six alerts and reminders for the physician. The reminders are selected by CHICA, using its Arden Syntax rule set based on the patient's EMR and answers provided on the tablet. Each alert has up to six check boxes with which the physician can document how s/he responded to the alert. The PWS, when completed, is scanned, the coded data corresponding to the check boxes are stored, and text is written into the physician's note in the medical record. CHICA may also produce any of a large number of handouts for helping the physician with assessment or patient education. CHICA also produces a summary of the patient's immunization history as well and advice on what shots the child is due to receive.

In an ongoing study of the Regenstrief-Merck collaboration, the investigators are studying the effect of providing physicians with a suggested "script" for recommending HPV vaccination to eligible patients' families. The study randomizes by physician whether the script is provided or whether the physician receives a simple reminder.

ELIGIBILITY:
Inclusion Criteria:

* Parents/legal guardians of 11-17 year old children.
* Children receive their healthcare at one of the 5 CHICA clinics.
* Parents are able to read either English or Spanish.
* Children have received no more than 2 doses of HPV vaccine

Exclusion Criteria:

* Parents will be excluded if their child is outside of the designated age range of 11-17 years, if the child has completed the 3-dose HPV vaccine series, or if the parent does not read either English or Spanish.

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1306 (Actual)
Dates: Start 2015-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Outcome Measure 1: Difference Between Average HPV Vaccine Series Initiation and Completion Rates | Seven Months
  Difference between average HPV vaccine series initiation and completion rates (as recorded in the CHIRP immunization registry) between sites using THEO integrated technology product compared to HPV Vaccination rates at Eskenazi sites not using THEO integrated technology product. Note that CHICA operates in 5 clinics in the Eskenazi Health Network. These clinics have been matched into two groups, each with 2 clinics, based on race and ethnicity of their patients. We will randomly assign one of these two groups to use THEO. The other group plus an additional CHICA clinic will continue to use CHICA without THEO.

SECONDARY OUTCOMES:
Outcome Measure 1: Relative Difference in Time of Appointment | Seven Months
  Relative differences in overall time of appointment for patient visits in which any dose of the HPV vaccine was given after using the integrated digital intervention, compared to overall time of appointment for patient visits in which any dose of the HPV vaccine was given after not using the integrated digital intervention

CONTACTS AND LOCATIONS:
Overall Officials: Gregory D Zimet, PhD, Principal Investigator — 317-274-8812
Locations (5):
- United States (5):
  - Eskenazi Health Outpatient Care Center, Indianapolis, Indiana
  - Eskenazi Health Center Blackburn, Indianapolis, Indiana
  - Eskenazi Health Center Forest Manor, Indianapolis, Indiana
  - Eskenazi Health West 38th Street, Indianapolis, Indiana
  - Eskenazi Health Pecar, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No
Individual provider data will not be shared.

REFERENCES:
- [Background] Parkin DM, Bray F. Chapter 2: The burden of HPV-related cancers. Vaccine. 2006 Aug 31;24 Suppl 3:S3/11-25. doi: 10.1016/j.vaccine.2006.05.111. PMID 16949997
- [Background] Giuliano AR, Anic G, Nyitray AG. Epidemiology and pathology of HPV disease in males. Gynecol Oncol. 2010 May;117(2 Suppl):S15-9. doi: 10.1016/j.ygyno.2010.01.026. Epub 2010 Feb 6. PMID 20138345
- [Background] Chaturvedi AK. Beyond cervical cancer: burden of other HPV-related cancers among men and women. J Adolesc Health. 2010 Apr;46(4 Suppl):S20-6. doi: 10.1016/j.jadohealth.2010.01.016. PMID 20307840
- [Background] Haupt RM, Sings HL. The efficacy and safety of the quadrivalent human papillomavirus 6/11/16/18 vaccine gardasil. J Adolesc Health. 2011 Nov;49(5):467-75. doi: 10.1016/j.jadohealth.2011.07.003. Epub 2011 Sep 9. PMID 22018560
- [Background] Arnheim-Dahlstrom L, Pasternak B, Svanstrom H, Sparen P, Hviid A. Autoimmune, neurological, and venous thromboembolic adverse events after immunisation of adolescent girls with quadrivalent human papillomavirus vaccine in Denmark and Sweden: cohort study. BMJ. 2013 Oct 9;347:f5906. doi: 10.1136/bmj.f5906. PMID 24108159
- [Background] Scheller NM, Svanstrom H, Pasternak B, Arnheim-Dahlstrom L, Sundstrom K, Fink K, Hviid A. Quadrivalent HPV vaccination and risk of multiple sclerosis and other demyelinating diseases of the central nervous system. JAMA. 2015 Jan 6;313(1):54-61. doi: 10.1001/jama.2014.16946. PMID 25562266
- [Background] Ojha RP, Jackson BE, Tota JE, Offutt-Powell TN, Singh KP, Bae S. Guillain-Barre syndrome following quadrivalent human papillomavirus vaccination among vaccine-eligible individuals in the United States. Hum Vaccin Immunother. 2014;10(1):232-7. doi: 10.4161/hv.26292. Epub 2013 Sep 6. PMID 24013368
- [Background] Klein NP, Hansen J, Chao C, Velicer C, Emery M, Slezak J, Lewis N, Deosaransingh K, Sy L, Ackerson B, Cheetham TC, Liaw KL, Takhar H, Jacobsen SJ. Safety of quadrivalent human papillomavirus vaccine administered routinely to females. Arch Pediatr Adolesc Med. 2012 Dec;166(12):1140-8. doi: 10.1001/archpediatrics.2012.1451. PMID 23027469
- [Background] Pedersen C, Petaja T, Strauss G, Rumke HC, Poder A, Richardus JH, Spiessens B, Descamps D, Hardt K, Lehtinen M, Dubin G; HPV Vaccine Adolescent Study Investigators Network. Immunization of early adolescent females with human papillomavirus type 16 and 18 L1 virus-like particle vaccine containing AS04 adjuvant. J Adolesc Health. 2007 Jun;40(6):564-71. doi: 10.1016/j.jadohealth.2007.02.015. PMID 17531764
- [Background] Reisinger KS, Block SL, Lazcano-Ponce E, Samakoses R, Esser MT, Erick J, Puchalski D, Giacoletti KE, Sings HL, Lukac S, Alvarez FB, Barr E. Safety and persistent immunogenicity of a quadrivalent human papillomavirus types 6, 11, 16, 18 L1 virus-like particle vaccine in preadolescents and adolescents: a randomized controlled trial. Pediatr Infect Dis J. 2007 Mar;26(3):201-9. doi: 10.1097/01.inf.0000253970.29190.5a. PMID 17484215
- [Background] Baandrup L, Blomberg M, Dehlendorff C, Sand C, Andersen KK, Kjaer SK. Significant decrease in the incidence of genital warts in young Danish women after implementation of a national human papillomavirus vaccination program. Sex Transm Dis. 2013 Feb;40(2):130-5. doi: 10.1097/OLQ.0b013e31827bd66b. PMID 23324976
- [Background] Ali H, Donovan B, Wand H, Read TR, Regan DG, Grulich AE, Fairley CK, Guy RJ. Genital warts in young Australians five years into national human papillomavirus vaccination programme: national surveillance data. BMJ. 2013 Apr 18;346:f2032. doi: 10.1136/bmj.f2032. PMID 23599298
- [Background] Ali H, Guy RJ, Wand H, Read TR, Regan DG, Grulich AE, Fairley CK, Donovan B. Decline in in-patient treatments of genital warts among young Australians following the national HPV vaccination program. BMC Infect Dis. 2013 Mar 18;13:140. doi: 10.1186/1471-2334-13-140. PMID 23506489
- [Background] Elam-Evans LD, Yankey D, Jeyarajah J, Singleton JA, Curtis RC, MacNeil J, Hariri S; Immunization Services Division, National Center for Immunization and Respiratory Diseases; Centers for Disease Control and Prevention (CDC). National, regional, state, and selected local area vaccination coverage among adolescents aged 13-17 years--United States, 2013. MMWR Morb Mortal Wkly Rep. 2014 Jul 25;63(29):625-33. PMID 25055186
- [Background] Brewer NT, Gottlieb SL, Reiter PL, McRee AL, Liddon N, Markowitz L, Smith JS. Longitudinal predictors of human papillomavirus vaccine initiation among adolescent girls in a high-risk geographic area. Sex Transm Dis. 2011 Mar;38(3):197-204. doi: 10.1097/OLQ.0b013e3181f12dbf. PMID 20838362
- [Background] Donahue KL, Stupiansky NW, Alexander AB, Zimet GD. Acceptability of the human papillomavirus vaccine and reasons for non-vaccination among parents of adolescent sons. Vaccine. 2014 Jun 30;32(31):3883-5. doi: 10.1016/j.vaccine.2014.05.035. Epub 2014 May 18. PMID 24844150
- [Background] Kester LM, Zimet GD, Fortenberry JD, Kahn JA, Shew ML. A national study of HPV vaccination of adolescent girls: rates, predictors, and reasons for non-vaccination. Matern Child Health J. 2013 Jul;17(5):879-85. doi: 10.1007/s10995-012-1066-z. PMID 22729660
- [Background] Holman DM, Benard V, Roland KB, Watson M, Liddon N, Stokley S. Barriers to human papillomavirus vaccination among US adolescents: a systematic review of the literature. JAMA Pediatr. 2014 Jan;168(1):76-82. doi: 10.1001/jamapediatrics.2013.2752. PMID 24276343
- [Background] Guerry SL, De Rosa CJ, Markowitz LE, Walker S, Liddon N, Kerndt PR, Gottlieb SL. Human papillomavirus vaccine initiation among adolescent girls in high-risk communities. Vaccine. 2011 Mar 9;29(12):2235-41. doi: 10.1016/j.vaccine.2011.01.052. Epub 2011 Feb 1. PMID 21288799
- [Background] Fu LY, Bonhomme LA, Cooper SC, Joseph JG, Zimet GD. Educational interventions to increase HPV vaccination acceptance: a systematic review. Vaccine. 2014 Apr 7;32(17):1901-20. doi: 10.1016/j.vaccine.2014.01.091. Epub 2014 Feb 14. PMID 24530401
- [Background] Kreuter MW, Strecher VJ, Glassman B. One size does not fit all: the case for tailoring print materials. Ann Behav Med. 1999 Fall;21(4):276-83. doi: 10.1007/BF02895958. PMID 10721433
- [Background] Lustria ML, Noar SM, Cortese J, Van Stee SK, Glueckauf RL, Lee J. A meta-analysis of web-delivered tailored health behavior change interventions. J Health Commun. 2013;18(9):1039-69. doi: 10.1080/10810730.2013.768727. Epub 2013 Jun 10. PMID 23750972
- [Background] Noar SM, Benac CN, Harris MS. Does tailoring matter? Meta-analytic review of tailored print health behavior change interventions. Psychol Bull. 2007 Jul;133(4):673-93. doi: 10.1037/0033-2909.133.4.673. PMID 17592961
- [Background] Gerend MA, Shepherd MA, Lustria ML. Increasing human papillomavirus vaccine acceptability by tailoring messages to young adult women's perceived barriers. Sex Transm Dis. 2013 May;40(5):401-5. doi: 10.1097/OLQ.0b013e318283c8a8. PMID 23588130
- [Background] Petty RE, Wegener DT, Fabrigar LR. Attitudes and attitude change. Annu Rev Psychol. 1997;48:609-47. doi: 10.1146/annurev.psych.48.1.609. PMID 9046570
- [Background] Carroll AE, Bauer NS, Dugan TM, Anand V, Saha C, Downs SM. Use of a computerized decision aid for ADHD diagnosis: a randomized controlled trial. Pediatrics. 2013 Sep;132(3):e623-9. doi: 10.1542/peds.2013-0933. Epub 2013 Aug 19. PMID 23958768
- [Background] Carroll AE, Biondich P, Anand V, Dugan TM, Downs SM. A randomized controlled trial of screening for maternal depression with a clinical decision support system. J Am Med Inform Assoc. 2013 Mar-Apr;20(2):311-6. doi: 10.1136/amiajnl-2011-000682. Epub 2012 Jun 28. PMID 22744960
- [Background] Carroll AE, Biondich PG, Anand V, Dugan TM, Sheley ME, Xu SZ, Downs SM. Targeted screening for pediatric conditions with the CHICA system. J Am Med Inform Assoc. 2011 Jul-Aug;18(4):485-90. doi: 10.1136/amiajnl-2011-000088. PMID 21672910
- [Background] Anand V, Carroll AE, Downs SM. Automated primary care screening in pediatric waiting rooms. Pediatrics. 2012 May;129(5):e1275-81. doi: 10.1542/peds.2011-2875. Epub 2012 Apr 16. PMID 22508925
- [Background] Biondich PG, Downs SM, Anand V, Carroll AE. Automating the recognition and prioritization of needed preventive services: early results from the CHICA system. AMIA Annu Symp Proc. 2005;2005:51-5. PMID 16779000
- [Background] Downs SM, Uner H. Expected value prioritization of prompts and reminders. Proc AMIA Symp. 2002:215-9. PMID 12463818
- [Background] Downs SM, Zhu V, Anand V, Biondich PG, Carroll AE. The CHICA smoking cessation system. AMIA Annu Symp Proc. 2008 Nov 6;2008:166-70. PMID 18998823
- [Derived] Dixon BE, Zimet GD, Xiao S, Tu W, Lindsay B, Church A, Downs SM. An Educational Intervention to Improve HPV Vaccination: A Cluster Randomized Trial. Pediatrics. 2019 Jan;143(1):e20181457. doi: 10.1542/peds.2018-1457. Epub 2018 Dec 10. PMID 30530637